CLINICAL TRIAL: NCT05015140
Title: Effects of Music Therapy on Sleep Quality in Patients Who Had Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sumeyye Can, Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HSCT
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hematologic Diseases
Keywords: hematopoietic stem cell transplant, music therapy, sleep quality
MeSH Terms: conditions — Hematologic Diseases; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): The first day before the application of music to each of the 15 patients in the experimental group (D-1) 'Patient Identification First evaluation will be made by filling the form "and then the" Richard Campbell Sleep Questionnaire ". The day before transplant (D-1) Starting from 10 days, calm music including nature sounds determined by the music therapist will be played using mp3 player. The Richard Campbell Sleep questionnaire will be filled again on the 10th day (D + 10) after the transplant.
  Interventions: Other: musıc therapy
- control group (No Intervention): - The day before the transplant (D-1) for each of the 15 patients in the control group, first 'Patient Identification Form' and then 'Richard The first evaluations will be made by filling the Campbell Sleep Questionnaire, and standard treatment and care interventions will be given to the patients in this group.
  The sleep questionnaire was filled out again on the tenth day (D + 10) after the transplant without any intervention.

INTERVENTIONS:
Other: musıc therapy — calm music with nature sounds set by the music therapist
  Arms: experiment group

SUMMARY:
In patients undergoing hematopoietic stem cell transplant; Side effects associated with high-dose chemotherapy and radiotherapy, night treatment and care, social isolation cause emotional problems and deterioration in sleep quality in this patient population. In a meta-analysis conducted in 2014, it was reported that music can be effective in improving sleep quality.

In this study, an experimental design with pre-test - post-test control group will be used to evaluate the effect of music therapy on sleep quality given to patients undergoing hematopoietic stem cell transplantation. It will be held between December 2020 and May 2021 at the Bone Marrow Transplantation Unit of Istanbul University-Cerrahpaşa Cerrahpaşa Medical Faculty Hospital. The population of the study will be the patients hospitalized in the unit within the specified date range and the sample number was determined as 30.

DETAILED DESCRIPTION:
Research Universe and Sample:

The population of the study will be the patients who applied to the Bone Marrow Transplantation Unit of Istanbul University-Cerrahpaşa Cerrahpaşa Medical Faculty Hospital between December 2020 - May 2021 and accepted the study. Considering the previous years in the date range of the study, it is predicted that an average of 25 patients will be hospitalized for stem cell transplantation. In a study conducted in 2014, it was reported that sleep disturbance continued in the long term after the transplantation in half of the patients who underwent hematopoietic stem cell transplantation. In the light of this information, the sample size was calculated as 24 using the OpenEpi program. Considering the possibility of patient or treatment-related disruptions during the study, it was planned to include 30 patients, 15 of which were experimental and 15 were control group.

Data Collection Tools The age, gender, type of transplant, habits and sleep of the patients created by the researcher during the data collection phase.

The "Patient Identification Form", which consists of 14 questions related to patients such as problems, and developed by Richards in 1987, was developed by Karaman Özlü et al. "Richard Campbell Sleep Questionnaire", whose validity and reliability study has been made, will be used.

Musical Intervention

In determining the music to be used, a quiet music containing the sounds of nature was determined in consultation with the music therapist.

It will be applied to the experimental group by using an mp3 player in the patient room, starting on the day before the transfer (D-1), every evening for 10 days and each session for 30 minutes. It will be applied between 23:00 and 24:00 in the evening so as not to prevent the standard treatment and care of the patients. After 10 days, the sleep quality of the patients will be re-evaluated using the Richard Campbell Sleep Questionnaire.

ELIGIBILITY:
Inclusion criteria in the study;

* To be conscious
* hospitalization for hematopoietic stem cell transplantation

Exclusion criteria;

* Deaf
* Terminal period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Richard Campbell Sleep Questionnaire | 10 days
  Evaluation of the change in sleep quality from baseline with the Richard Campbell sleep questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul
  - İstanbul University- Cerrahpaşa, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided